CLINICAL TRIAL: NCT02119221
Title: Single Center, Open-label, Non-randomized, Non-placebo-controlled Study to Investigate the Metabolism, Excretion Pattern, Mass Balance, Safety, Tolerability and Pharmacokinetics After Single Intravenous Administration of 12 mg [14C]Copanlisib (BAY 80-6946) in Healthy Male Subjects
Brief Title: Copanlisib Mass Balance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16353; 2013-002544-90 (EudraCT Number)
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]Copanlisib (Experimental)
  Interventions: Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (BAY80-6946) — Intravenous infusion of 12 mg copanlisib labeled with 2.76 MBq (75 μCi) of [14C]

SUMMARY:
The study aims to provide understanding of the relative relevance of the different excretion pathways of Copanlisib in humans, as well as to characterize its metabolite profile.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 45 to 65 years
* Body weight greater or equal to 60 kg and body mass index (BMI): above/equal 18 and below/equal 30 kg/m²

Exclusion Criteria:

* Regular use of medicines
* Known recent (last 2 years) abuse of recreational drugs, suspicion of drug or alcohol abuse, or positive results of the drug and alcohol screen tests at screening or baseline
* Use of strong inhibitors of cytochrome P450 (CYP)3A4, as well as use of St John's Wort or strong inducers of CYP3A4 prohibited from 14 days before the administration of study drug until discharge from the clinic
* Smoking
* Average intake of more than 24 units of alcohol per week; Regular daily consumption of more than 1 L of methylxanthine-containing beverages
* Any condition, which may result in longer than usual retention of urine or feces in the body, such as pronounced (less than one defecation in 2 days) constipation or symptomatic prostatic hypertrophy.
* Participation in another mass balance study with a radiation burden > 0.1 mSv in the period of 1 year before screening

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of copanlisib in plasma by maximum concentration (Cmax) | Multiple time points up to 336 hours
Pharmacokinetics of copanlisib in plasma by area under the measured matrix concentration versus time curve from the first time point (t=0) extrapolated to infinity (AUC) | Multiple time points up to 336 hours
Pharmacokinetics of copanlisib in plasma by area under the measured matrix concentration versus time curve to the last data point above the lower limit of quantitation (AUC(0-tlast)) | Multiple time points up to 336 hours
Pharmacokinetics of total radioactivity in plasma by Cmax | Multiple time points up to 336 hours
Pharmacokinetics of total radioactivity in plasma by AUC | Multiple time points up to 336 hours
Pharmacokinetics of total radioactivity in plasma by AUC(0-tlast) | Multiple time points up to 336 hours
Pharmacokinetics of total radioactivity in whole blood by Cmax | Multiple time points up to 336 hours
Pharmacokinetics of total radioactivity in whole blood by AUC | Multiple time points up to 336 hours
Pharmacokinetics of total radioactivity in whole blood by AUC(0-tlast) | Multiple time points up to 336 hours
Radioactivity excreted in urine as a percentage of the dose (AE,ur) | Multiple time points up to 336 hours
Radioactivity excreted in feces as a percentage of the dose (AE,fec) | Multiple time points up to 336 hours
Metabolite profile in plasma | Multiple time points up to 336 hours
Metabolite profile in urine | Multiple time points up to 336 hours
Metabolite profile in feces | Multiple time points up to 336 hours

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Until 30 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Zuidlaren, Netherlands